CLINICAL TRIAL: NCT00942786
Title: Prospective Study to Evaluate the Predictive Value of Brain Natriuretic Peptides for Adverse Long-term Cardiac Outcome
Brief Title: Natriuretic Peptides - Predictors of In-hospital and Long-term Major Adverse Cardiac Events After Emergency Surgery?
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 19-077 ex 07/08
Record Dates: First submitted 2009-07-18; First posted 2009-07-21 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Surgery
Keywords: natriuretic peptides; emergency non-cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — one vial of serum per patient is retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: Consecutive patients undergoing emergency surgery

SUMMARY:
The investigators hypothesize that the level of perioperative natriuretic peptides is associated with in-hospital and long term major adverse cardiac events.

DETAILED DESCRIPTION:
The purpose of the study is to measure levels of brain natriuretic peptides before and after urgent non-cardiac surgery and to evaluate their predictive value for adverse long-term outcome.

ELIGIBILITY:
Inclusion criteria:

* Emergency surgery:

  1. Vascular
  2. Intra-abdominal
  3. Orthopedic

     Exclusion Criteria:
* Patients unable to provide informed consent
* Thoracic surgery
* Trauma surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing emergency non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2008-02; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Mahla, M.D., Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Medical University of Graz
Locations (1):
- Department of Anesthesia and Intensive Care Medicine, Graz, Austria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Treatment
Started | 297
Completed | 297 (date of last follow-up)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- One Arm: consecutive patients presenting for emergent non-cardiac surgery
Arm/Group | One Arm
Number analyzed (Participants) | 297
Age, Continuous [Mean (Full Range); unit: years] | 74 [51 to 103]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 117

OUTCOME MEASURES:

1. Primary Outcome: Occurence of Adverse Cardiac Events
Description: Occurence of major adverse cardiac events (composite of nonfatal myocardial infarction, acute heart failure or death).
  Non-fatal Myocardial infarction was defined as a typical increase and decrease of troponin together with evidence of myocardial ischemia with at least one of the following: symptoms of ischemia, ECG changes indicative of ischemia or new Q waves, or imaging evidence of new regional wall motion abnormality.
  Acute heart failure was defined as clinical signs and symptoms of heart failure with echocardiographic evidence of cardiac dysfunction and clinical response to treatment directed towards heart failure.
Time Frame: postoperatively (index surgery) until a median follow-up of 34 months
Measure: Number; unit: participants
Arm/Group | No Treatment
Number analyzed (Participants) | 297
participants | 91

2. Other Pre Specified Outcome: NT-ProBNP Preoperative
Description: NT-ProBNP was measured 0-24 hours before induction of anesthesia
Time Frame: 0-24 hours before induction of anesthesia
Population: Consecutive patients undergoing emergent non-cardiac surgery
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- All Patients: Consecutive patients undergoing emergent non-cardiac surgery
Arm/Group | All Patients
Number analyzed (Participants) | 297
pg/ml | 491 [189 to 1670]

3. Other Pre Specified Outcome: Association Between Preoperative NT-ProBNP and Occurence of Adverse Cardiac Events
Description: Evaluation of the association between preoperative NT-ProBNP and occurence of adverse cardiac events
Time Frame: postoperatively (index surgery) until a median follow-up of 34 months
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Patients Sustaining Adverse Events: Subjects who reached the primary endpoint
- Patients Not Sustaining Adverse Events: Subjects who did not reach the primary endpoint
Arm/Group | Patients Sustaining Adverse Events | Patients Not Sustaining Adverse Events
Number analyzed (Participants) | 91 | 206
pg/ml | 1527 [544 to 3650] | 296 [119 to 873]

ADVERSE EVENTS:
Time Frame: Median follow-up of 34 months
Groups:
- One Arm: consecutive patients presenting for emergent non-cardiac surgery
  Patients were followed for occurence of major adverse cardiac events
Arm/Group | One Arm
Serious Adverse Events (participants affected / at risk) | 91/297
Other Adverse Events (participants affected / at risk) | 0/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Arm (N=297)
Serious Adverse cardiac events (Cardiac disorders) | 91 (91)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes